CLINICAL TRIAL: NCT04207996
Title: High Resolution, Noninvasive Measurement and Functional Classification of Vagal Nerve Response Patterns in Relation to Gastroparesis Symptom Management Using Gastric Electrical Stimulation Therapy
Brief Title: Vagus Nerve Response in Gastroparesis Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Purdue University (Other)
Responsible Party: Principal Investigator, Thomas V. Nowak, Clinical Professor and Principal Investigator, Indiana University
Other Study IDs: MEA study
Record Dates: First submitted 2019-12-17; First posted 2019-12-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to characterize how vagus nerve compound action potentials (CNAPs) conduct along the vagus nerve in gastroparetic patients receiving GES therapy using a flexible, non-invasive multielectrode array (MEA).

DETAILED DESCRIPTION:
During Phase

1, in a small cohort of 5-10 gastroparetic patients receiving GES therapy, we will determine the optimal multielectrode array (MEA) recording electrode configuration (e.g., surface area covered and electrode density) for the noninvasive measurement of gastric electrical stimulation (GES) evoked compound nerve action potentials (CNAP) from the skin surface over the left and right cervical vagus nerve. During Phase 2, a study of 15-30 gastroparetic patients receiving GES therapy, we will use the optimal MEA configuration identified in Task 1 to measure and classify the vagal CNAP response signature (including the direction of travel and anatomical location of the strongest signal (e.g., to infer the anatomical course of the cervical vagus in each subject) with respect to subject-reported symptom scores via the 9-item Gastroparesis Cardinal Symptom Index (GCSI) survey. We will cross-reference these results with the preliminary results obtained with bipolar ECG electrodes.

Phase 1:

Subjects will complete a symptom survey questionnaire and Gastric Cardinal Symptom Index (GCSI) questionnaire. Two electrocardiography (ECG) electrodes will be placed on both sides of the neck overlying the area near the carotid pulse (which overlies the carotid artery in the neck on the side of your neck) where the vagus nerve is located.This is done in order to measure the vagal nerve electrical impulses in the neck (electrical signal travelling in the nerve).

Two ECG electrodes will be placed on each of the arms and one on the chest for measurement of electrocardiogram (ECG) ( a test to measure the electrical activity of your heart). Three ECG electrodes may be placed on the stomach to measure the electrical activity of the stomach.

After the placement of the electrodes, a 2-5 minute recording will be made.The GES device will be interrogated (data will be obtained) for the settings of the device and these will be recorded by the study team. After the recording, the electrodes will be removed from the neck and a newer kind of electrodes called as MEA (Multi electrode Array)) devices that contain multiple (tens to thousands of small electrodes) will be placed on either one, or both sides of the neck. This film will help capture the vagus signal from a large area and help define the path of the vagus nerve. After the placement of this film with small electrodes, another 2-5 minute recording will be made. The electrodes will then be removed and subject will be allowed to go home.

The total time required for Phase 1 will be approximately an hour (60 minutes).

Phase 2:

Subject will complete a symptom survey questionnaire and Gastric Cardinal Symptom Index (GCSI) questionnaire. Multiple electrodes (MEA) will be placed on either one or both sides of the neck. One ECG electrodes will be placed on each of the arms, and one on the chest for measurement of electrocardiogram (ECG). Three ECG electrodes will be placed on the stomach to measure the electrical activity of the stomach. After the placement of the electrodes a 2-5 minute recording will be made. The GES device will be interrogated (data will be obtained) for the settings and these will be recorded by the study team. With the GES stimulator on, a 2-5 minute recording will be made. Then, the GES stimulator will be reprogrammed to deliver the signal at 50% of the original power, and another 2-5 minute recording will be made. Then, the device will again be programmed to deliver the signal at 25% of the original power setting on the device. Another 2-5 minute recording will be made. After this, the device will be reprogrammed to the original settings. The electrodes will then be removed and subject will be allowed to go home.

The total time required for Phase 2 will be approximately an hour (60 minutes).

ELIGIBILITY:
Inclusion Criteria:

1. Gastroparetic patient with a stimulator (Enterra Device placed)
2. Aged 18-80 years
3. Willing to have electrodes placed on the neck

Exclusion Criteria:

1. Unable to provide consent
2. Pregnant females
3. Prisoners

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects 18 years and above who have a gastric electrical stimulator placed for gastroparesis
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Optimal MEA configuration | 3 years
  Identify the optimal MEA configuration for vagal response capture
GES and symptom survey | 3 years
  Identify the compound nerve action potential in each subject and correlate that with the symptom survey data collected for each subject

CONTACTS AND LOCATIONS:
Overall Officials: Thomas V Nowak, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Hosptial, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT04207996/ICF_000.pdf